CLINICAL TRIAL: NCT06839872
Title: BOSS: BTK Inhibitor Optimal Sequencing Study Phase II Open-label Single Arm Trial of Pirtobrutinib in Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma After First-line Acalabrutinib Progression
Brief Title: A Study to Investigate the Sequencing Strategy of Pirtobrutinib After Disease Progression on First-line Acalabrutinib Treatment for Adult Participants With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Acronym: BOSS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: AstraZeneca has made the decision to cancel the trial.
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8220R00065
Record Dates: First submitted 2025-01-21; First posted 2025-02-21 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — pirtobrutinib; acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pirtobrutinib and Acalabrutinib (Experimental): Participants will receive dose A of pirtobrutinib starting Cycle 1 Day 1 for up to 24 cycles or until disease progression, unacceptable toxicity, death, or withdrawal of consent. If they progress on pirtobrutinib, a subset will receive dose B of acalabrutinib starting Cycle 1 Day 1 for up to 12 cycles or until disease progression, death, intolerance, unacceptable toxicity, or withdrawal of consent. Those benefiting from treatment will enter the Disease Follow-up period, continuing with pirtobrutinib or acalabrutinib until disease progression, unacceptable toxicity, death, or withdrawal of consent. After 36 months from starting pirtobrutinib, participants can continue receiving treatment off-trial if beneficial, in consultation with their physician.
  Interventions: Drug: Pirtobrutinib; Drug: Acalabrutinib

INTERVENTIONS:
Drug: Pirtobrutinib — Patients will receive pirtobrutinib orally with dosing schedule as prescribed
  Other Names: JAYPIRCA
Drug: Acalabrutinib — Patients will receive acalabrutinib orally with dosing schedule as prescribed.
  Other Names: CALQUENCE®

SUMMARY:
To assess the efficacy and safety of pirtobrutinib in participants with CLL/SLL who have progressed on first-line treatment with acalabrutinib.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy and safety of pirtobrutinib in participants with CLL/SLL who have progressed on first-line treatment with acalabrutinib. A subset of participants who have disease progression on pirtobrutinib will be retreated with acalabrutinib to assess whether relapsed CLL can be re-sensitized to a covalent irreversible BTK inhibitor such as acalabrutinib, and thereby, remain on treatment within the BTK inhibitor class rather than transition into another CLL/SLL treatment.

* The study duration for each participant will be up to 3 years in total.
* For participants who receive pirtobrutinib alone, the visit frequency will be approximately every month for the first 6 months. After that, the visit frequency will be reduced to one visit approximately every 3 months for the subsequent 12 months. The final part of the Treatment Phase has 2 visits in the space of 6 months. There is one visit to the site after the Treatment Phase.
* Participants who have disease progression on pirtobrutinib and go on to receive acalabrutinib retreatment will visit the site approximately once every month for the first 6 months. After that, the visit frequency will be reduced to 2 visits in the space of 6 months. There is one visit to the site after the Treatment Phase.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 at the time of signing the informed consent.
* Participants must have received acalabrutinib monotherapy as first-line treatment for CLL/SLL, have progressed per the iwCLL Criteria (Hallek et al 2018) and be eligible for second-line treatment by the same criteria.
* ECOG performance status of 0, 1, or 2.
* Adequate organ and BM function.
* Adequate coagulation, defined as aPTT or PTT and PT or INR not greater than 1.5 × ULN.
* Participants have a clearly defined, documented and accessible start date of their first line acalabrutinib monotherapy for CLL/SLL.
* Participants are eligible for the acalabrutinib retreatment phase only if they have progressed on pirtobrutinib monotherapy per iwCLL Criteria.

Exclusion Criteria:

* Major surgical procedure within 30 days before and not recovered adequately the first dose of study drug.
* Participants who experienced a major bleeding event or Grade ≥ 3 arrhythmia on prior treatment with a BTK inhibitor.
* History of bleeding diathesis (eg, hemophilia, von Willebrand disease).
* History of stroke or intracranial hemorrhage within 6 months before first dose of study drug.
* Significant cardiovascular disease.
* History of PML.
* Any active significant infection.
* HIV positive
* Active HBV or HCV infection.
* Active CNS involvement by lymphoma, leptomeningeal disease, or spinal cord compression.
* Active auto-immune cytopenia.
* History of prior or current malignancy.
* Requires or receiving therapeutic anticoagulation with warfarin or equivalent vitamin K antagonists.
* Received a live virus vaccination within 28 days of first dose of study drug.
* Requires treatment with a strong CYP3A inhibitor or inducer. The use of strong CYP3A inhibitors within 1 week or strong CYP3A inducers within 3 weeks of the first dose of study drug is prohibited.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2028-07-28 (Estimated); Study Completion 2030-07-29 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) in participants with CLL/SLL. | ORR will be assessed after 12 cycles (each cycle lasts 28 days) of pirtobrutinib.
  ORR is defined as the proportion of participants who achieve best response of CR, CRi, nPR, or PR per the iwCLL Criteria as assessed by the investigator.

SECONDARY OUTCOMES:
Investigator assessed ORR in participants with CLL/SLL. | ORR will be assessed after 24 cycles (each cycle is 28 days) of pirtobrutinib and at 3 years from Cycle 1: Day 1 of pirtobrutinib.
  ORR is defined as the proportion of participants who achieve best response of CR, CRi, nPR, or PR per the iwCLL Criteria as assessed by the investigator.
Progression free Survival (PFS) in participants with CLL/SLL. | PFS will be assessed at 24 months of pirtobrutinib treatment.
  PFS is defined as time from date of the first dose of pirtobrutinib until disease progression per the iwCLL Criteria as assessed by the investigator, or death due to any cause in the absence of disease progression.
Safety and tolerability of pirtobrutinib in CLL/SLL following disease progression on first-line acalabrutinib in participants with CLL/SLL. | Safety and tolerability will be evaluated at every visit starting from pirtobrutinib treatment through the study completion (for 3 years)
  Safety and tolerability will be evaluated as the number of participants with Adverse Events (AEs), Serious Adverse Events (SAEs), and AE leading to treatment discontinuation.
Safety of acalabrutinib retreatment following disease progression on pirtobrutinib in participants with CLL/SLL. | Safety will be evaluated at every visit starting from acalabrutinib treatment through the study completion (for 3 years)
  Safety will be evaluated as the number of participants with Adverse Events (AEs), Serious Adverse Events (SAEs), and AE leading to treatment discontinuation.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/